CLINICAL TRIAL: NCT01083615
Title: A Randomized, Placebo-Controlled, Double-Blind, Phase 3 Study Evaluating the Pain Palliation Benefit of Adding Custirsen to a Taxane for Second-Line Chemotherapy in Men With Castrate Resistance Prostate Cancer
Brief Title: A Study Evaluating the Pain Palliation Benefit of Adding Custirsen to Docetaxel Retreatment or Cabazitaxel as Second Line Therapy in Men With Metastatic Castrate Resistant Prostate Cancer (mCRPC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to enroll due to criteria for stable baseline pain
Sponsor: Achieve Life Sciences (Industry)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OGX-011-10
Record Dates: First submitted 2010-02-26; First posted 2010-03-10 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Castrate-Resistant Prostate Cancer; Hormone Refractory Prostate Cancer
Keywords: CRPC patients with cancer related pain; CRPC; HRPC
MeSH Terms: interventions — OGX-011; Sodium Chloride; Docetaxel; cabazitaxel; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Custirsen (Experimental): Study treatment starts with a Loading Dose Period (1 week) during which 3 infusions of custirsen will be administered. Following the Loading Dose Period, study treatment will consist of docetaxel (75 mg/m2 total dose) or cabazitaxel (25 mg/m2 total dose) on a 21-day cycle with weekly custirsen infusions (640 mg total dose) on Day 1, 8 and 15 of each 21-day cycle and oral prednisone BID.
  Participants will continue study treatment until pain progression, unacceptable toxicity, completion of 10 cycles or other specific criteria for withdrawal identified in the protocol.
  Interventions: Drug: custirsen sodium; Drug: docetaxel; Drug: cabazitaxel; Drug: prednisone
- Placebo (Placebo Comparator): Study treatment starts with a Loading Dose Period (1 week) during which 3 infusions of placebo (isotonic, 0.9% sodium chloride) will be administered. Following the Loading Dose Period, study treatment will consist of docetaxel (75 mg/m2 total dose) or cabazitaxel (25 mg/m2 total dose) on a 21-day cycle with weekly placebo infusions on Day 1, 8 and 15 of each 21-day cycle and oral prednisone BID.
  Participants will continue study treatment until pain progression, unacceptable toxicity, completion of 10 cycles or other specific criteria for withdrawal identified in the protocol.
  Interventions: Drug: isotonic, 0.9% sodium chloride; Drug: docetaxel; Drug: cabazitaxel; Drug: prednisone

INTERVENTIONS:
Drug: custirsen sodium — An antisense oligonucleotide that blocks production of clusterin
  Other Names: OGX-011
  Arms: Custirsen
Drug: isotonic, 0.9% sodium chloride — Placebo for custirsen sodium
  Arms: Placebo
Drug: docetaxel
Drug: cabazitaxel
Drug: prednisone

SUMMARY:
The purpose of this study is to determine if the addition of study drug (custirsen) can provide durable pain palliation for castrate resistant prostate cancer patients receiving docetaxel retreatment or cabazitaxel as a second line therapy.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter, international trial enrolling patients with metastatic CRPC who had a response to first-line docetaxel therapy and have prostate cancer-related pain with progression of disease. The intended intervention is second-line treatment with docetaxel retreatment or cabazitaxel plus study agent, where custirsen is to be administered in the investigational arm and placebo is to be administered in the control arm.

Selection of the chemotherapy (docetaxel re-treatment or cabazitaxel) is to be determined by the treating physician, based on the patient's first-line response.

The study will primarily assess pain and analgesic use for evaluation of durable pain palliation in response to study treatment. Pain and analgesic use will be obtained via a 3rd party contact center (direct contact with patient).

Study treatment starts with a Loading Dose Period during which three infusions of study agent (custirsen vs. placebo) will be administered. Following the Loading Dose Period, study treatment will consist of docetaxel or cabazitaxel on a 21-day cycle with weekly study agent (custirsen vs. placebo) infusions on Day 1, 8 and 15 of each 21-day cycle and oral prednisone BID.

Patients will continue study treatment until pain progression, unacceptable toxicity, completion of 10 cycles or other specific criteria for withdrawal identified in the protocol. If study treatment is completed or discontinued prior to pain progression, 6-day assessments will continue every 3 weeks until pain progression is documented. Follow-up after study treatment will occur for safety parameters for 3 weeks after the last study agent infusion in all patients. Survival status updates are to be reported every 12 weeks following documentation of pain progression. The amount of time that patients remain on the study will vary; but the average survival of these patients who receive second line taxane treatment is expected to be 14 to 15 months.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years on the date of consent.
2. Histological or cytological diagnosis of adenocarcinoma of the prostate.
3. Metastatic disease at screening on a chest, abdomen or pelvic CT or bone scan.
4. Concurrent pain and analgesic use that is viewed by the Investigator to be related to prostate cancer.
5. Received at least 4 cycles of prior docetaxel-based first-line chemotherapy for metastatic disease based on a q3 week schedule of docetaxel. Patients treated on a weekly or alternate schedule for first-line docetaxel must have received an accumulated dose of docetaxel of at least 300 mg/M2.
6. Current progressive disease during or after completing first-line docetaxel treatment.
7. Baseline laboratory values at screening visit within protocol defined limits.
8. Must be willing to continue primary androgen suppression with luteinizing hormone releasing hormone (LHRH) analogues throughout the study, if not treated with bilateral orchiectomy.
9. Adequate bone marrow function.
10. Karnofsky score ≥ 70% at screening visit.
11. At least 21 days have passed since completing radiotherapy at the time of randomization.
12. At least 21 days have passed since completing any cytotoxic agent or investigational agent given in combination with the docetaxel-based first-line therapy, including ASOs (except custirsen which is an exclusion criterion), at the time of randomization.
13. Has recovered from all therapy related toxicity to ≤ grade 2 (except alopecia, anemia and any signs or symptoms of androgen deprivation therapy).
14. Patient can tolerate a starting dose of docetaxel of 75 mg/M2 or cabazitaxel at 25 mg/M2.
15. Patient must have remained on the same bisphosphonate or denosumab usage for a minimum of 12 weeks prior to randomization.
16. Written informed consent must be obtained prior to any protocol-specific procedures being performed.

Exclusion Criteria

1. More than two interruptions in first-line docetaxel therapy. An interruption will be defined as more than 6 weeks between doses.
2. Life expectancy less than 12 weeks.
3. Previously participated in any clinical trial evaluating custirsen.
4. Received any other cytotoxic chemotherapy as a second-line treatment after first-line docetaxel-based therapy.
5. Not on any opioid analgesic regimen for their prostate cancer-related pain.
6. Receiving more than one drug within each of the separate categories of long-acting opioid, short-acting opioid, and non-opioid.
7. Receiving any analgesic specified in the protocol as unacceptable for this study.
8. Planned concomitant participation in another clinical trial of an experimental agent, vaccine or device. Concomitant participation in observational studies is acceptable.
9. Inability to communicate and read in English, Spanish or French.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To ascertain whether the investigational arm has a greater proportion of patients with durable pain palliation as compared to the control arm. | 3 to 6 months

SECONDARY OUTCOMES:
To ascertain whether patients randomized to the investigational arm have a longer time to pain progression as compared to patients randomized to the control arm. | 6 months.
Safety | 6 months
  Comparison of treatment arms with respect to the incidence of serious adverse events and the incidence of grade 3 or higher adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz M Beer, M.D., Principal Investigator — Oregon Health and Science University; Sebastien J Hotte, M.D., Principal Investigator — Juravinski Cancer Centre, McMaster University; Karim Fizazi, M.D., Ph.D., Principal Investigator — Institut Gustave Roussy, University of Paris
Locations (33):
- United States (20):
  - La Verne, California
  - Fort Lauderdale, Florida
  - Tampa, Florida
  - Honolulu, Hawaii
  - Urbana, Illinois
  - Metairie, Louisiana
  - Baltimore, Maryland
  - Burlington, Massachusetts
  - Detroit, Michigan
  - Kansas City, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Syracuse, New York
  - Raleigh, North Carolina
  - Canton, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Columbia, South Carolina
  - Memphis, Tennessee
  - Tyler, Texas
- Canada (2):
  - Winnipeg, Manitoba
  - Hamilton, Ontario
- France (4):
  - Lyon
  - Paris
  - Saint-Herblain
  - Villejuif
- Spain (5):
  - Barcelona
  - Madrid
  - Pamplona
  - Sabadell
  - Valencia
- United Kingdom (2):
  - Cambridge
  - Sutton